CLINICAL TRIAL: NCT07011381
Title: Parental Perception of Oral Health-Related Quality of Life Among Sudanese Refugee Children Compered to Egyptian Children
Brief Title: Parental Perception of Oral Health-Related Quality of Life in Sudanese Refugee vs. Egyptian Children
Status: Enrolling by invitation | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, SHOGI BOREY ELBOSHRA SULIAMAN, Principal Investigator, Kafrelsheikh University
Other Study IDs: KFSIRB200-599
Record Dates: First submitted 2025-05-09; First posted 2025-06-08 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Dental Caries; Gingivitis; Oral Health; Refugee Health
Keywords: dental caries; gingivitis; oral health; refugee health
MeSH Terms: conditions — Dental Caries; Gingivitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sudanese Refugee Children Group: Children aged 6-12 years residing in [location], identified as Sudanese refugees. Participants will undergo clinical oral health assessment and complete a child oral health quality of life questionnaire (COHIP). Parental perception will be documented through structured interviews.
- Egyptian Children Group: Children aged 6-12 years residing in [location], identified as native Egyptian citizens. Participants will undergo clinical oral health assessment and complete the same COHIP questionnaire. Parental perception will also be recorded via interviews.

SUMMARY:
This cross-sectional analytical study aims to assess and compare parental perceptions of oral health-related quality of life (OHRQoL) among Sudanese refugee children and Egyptian children aged 6-12 years living in Egypt. The study will include 192 child-parent pairs (96 Sudanese refugees and 96 Egyptians). Data will be collected via a validated Arabic questionnaire adapted from the Child Oral Health Impact Profile (COHIP) and clinical oral health examinations using DMFT/dmft indices, Gingival Index, and Plaque Index. The study seeks to identify disparities in oral health, parental awareness, and access to dental care services, thereby informing future community-based interventions and public health policies targeting vulnerable populations such as refugee children.

ELIGIBILITY:
Inclusion Criteria:

Children aged 6-12 years

Either Sudanese refugee or Egyptian national

Resident in Cairo for at least 1 year

Informed consent obtained from parent or legal guardian

Exclusion Criteria:

Systemic health conditions affecting oral health

Ongoing orthodontic treatment

Children with special health care needs or developmental disabilities

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Sudanese refugee and Egyptian children aged 6-12 years attending selected schools and community centers in Cairo, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Mean Total Score on the Child Oral Health Impact Profile (COHIP) Questionnaire | Baseline (single clinical visit at enrollment)
  Measured using the validated Arabic version of the Child Oral Health Impact Profile (COHIP) questionnaire. Total score and domain-specific subscores (Oral Health, Functional Well-being, Emotional Well-being, School Environment, and Self-image) will be analyzed.
  Full name: Child Oral Health Impact Profile (COHIP), Arabic version
  Score range: 0 to 140
  Higher scores = better oral health-related quality of life

SECONDARY OUTCOMES:
Clinical Oral Health Status | Baseline (Day 1, clinical oral examination)
  Includes the DMFT/dmft index (Decayed, Missing, and Filled Teeth), plaque index, and gingival index, assessed by calibrated dental examiners according to WHO guidelines.
  Outcome 1 : Mean Decayed, Missing, and Filled Teeth (DMFT/dmft) Index Score
  Unit: index score (range 0-28 or appropriate scale)
  Outcome 2 : Mean Plaque Index Score
  Unit: index score ( 0-3)
  Outcome 3 : Mean Gingival Index Score
  Unit: index score ( 0-3)

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Faculty of Oral and Dental Medicine, Kafr ash Shaykh, Kafr Ash Shaikh/ Elhamrawy, Egypt

IPD SHARING:
Plan to Share IPD: No